CLINICAL TRIAL: NCT05179499
Title: Early Vasopressors in Sepsis
Acronym: EVIS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Edinburgh (Other); Northern Care Alliance NHS Foundation Trust (Other); University of Manchester (Other); University of Glasgow (Other); NHS Lothian (Other Government); Chelsea and Westminster NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GN20AE342; 2021-006886-39 (EudraCT Number)
Record Dates: First submitted 2021-11-11; First posted 2022-01-05 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Sepsis
Keywords: Sepsis; Resuscitation; Norepinephrine; Intravenous fluids; Emergency Medicine; Critical Care
MeSH Terms: conditions — Sepsis | interventions — Norepinephrine

STUDY DESIGN:
Intervention Model Description: Open label, two arm, multicentre, pragmatic parallel group randomised trial with an internal pilot
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Active Comparator): Participants will receive peripheral vasopressor infusion of norepinephrine (16 micrograms/ml) during the initial 48 hour study period. All other care will be as per local protocol.
  Interventions: Drug: Norepinephrine
- Standard care (Placebo Comparator): Participants allocated to the control arm will receive standard care as defined by the UK NICE guidelines and the Surviving Sepsis Campaign guidelines during the 48 hour study period post randomisation. All other care will be as per local protocol.
  Interventions: Other: Balanced Crystalloid

INTERVENTIONS:
Drug: Norepinephrine — Norepinepherine should be prepared and delivered at a concentration of 16 micrograms/ml
  Arms: Intervention Arm
Other: Balanced Crystalloid — IV fluids administered as per standard care
  Arms: Standard care

SUMMARY:
Sepsis is a life-threatening reaction to an infection. It happens when the immune system overreacts to an infection and starts to damage the body's tissues and organs.

The aim of this research study is to compare the two different ways to treat sepsis, in the early phase of treatment immediately after the participants arrive in hospital. The standard approach is to give a salt solution fluid through a drip in the participants arm to start with, then adding in a medication that increases the blood flow to the participants vital organs (a vasopressor mediation called norepinephrine) if required. The alternative approach is to start the vasopressor medication immediately, and then add in extra salt solution fluid via a drip if required. Vasopressors work by increasing the blood pressure which allows a better blood flow to the internal organs. The investigators plan to see which approach is better and to see if they have a role in improving a patient's recovery time, reducing complications, the length of time they stay in hospital and longer term poor health.

Based on research that has already been done, the investigators believe treating patients with vasopressors when they arrive in the Emergency Department, may have potential advantages over the standard fluids used today. However, the evidence is not clear and that is why this research is being done.

DETAILED DESCRIPTION:
Sepsis results from overwhelming reactions to microbial infections where the immune system initiates dysregulated responses that lead to remote organ dysfunction, shock and ultimately death. Sepsis remains a significant global issue - as well as direct mortality, survivors suffer long term reductions in patient centred outcomes, with reduced quality of life and functional status. Patients with hypotension and organ hypoperfusion as a result of sepsis have poorer outcomes by dysregulated inflammation, endothelial dysfunction, immune suppression, and organ dysfunction. Current guidelines highlight the importance of early fluid resuscitation, but the association of early fluid therapy with improved outcomes is unclear. In the resuscitation phase, current practice is to give intravenous (IV) fluid and intermittent vasopressor boluses if required, before, for some patients, continuous vasopressor infusion via a central venous line in Intensive Care (ICU). An alternative, early continuous peripheral vasopressor infusion (PVI) is not routine practice in the UK.

Current practice in the UK is guided by NICE Sepsis guidance and the international Surviving Sepsis Campaign (SSC) consensus recommendations. Both specify intravenous fluid administration as a central tenet of early resuscitation of patients with septic shock, with intravenous vasopressor administration recommended after intravenous fluid resuscitation. NICE recommend boluses of 500ml of crystalloid and "refer to critical care for review of management including need for central venous access and initiation of vasopressors". SSC recommend 30ml/kg crystalloid in first hour, followed by vasopressors to maintain MAP>65.

The current NICE fluid resuscitation guideline, November 2020, continues to emphasise 500ml boluses of crystalloid as usual care. A recent international survey of 100 critical care and EM physicians regarding intravenous fluid resuscitation practice, confirmed that an initial bolus of 1000ml of crystalloid, followed by 500ml boluses of crystalloid remained the most common management strategy for the initial treatment of septic shock. This persisted despite the lack of benefit demonstrated in three landmark trials of protocolised sepsis management.

In recent years, there has been increasing acceptance of peripheral administration of norepinephrine, based on evidence of safety and efficacy. The Intensive Care Society published guidance on peripheral vasopressor infusion in November 2020. We have recently conducted a survey amongst ED and ICU clinicians in the UK regarding attitudes and current practice related to the use of intravenous peripheral vasopressors. Eighty two respondents provided the following answers

1. Experience of use of any intravenous vasopressor in ED was high (81%);
2. Exclusive PVI made up 23% of all vasopressor use in ED;
3. Norepinephrine (norepinephrine) was the most common vasopressor (54%);
4. Barriers to PVI were local protocols and an appropriate level of care in the destination ward for a patient on vasopressor infusion.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Clinically suspected or proven infection resulting in principal reason for acute illness
* SBP < 90 mmHg or MAP of < 65 mmHg (within an hour of eligibility assessment)
* Measured serum lactate of > 2 mmol/L. The serum lactate should be measured 2 hours prior to determination of eligibility, where possible. Longer timeframes may be used and justified within the medical notes if, in the opinion of the investigator, the clinical status of the patient has not significantly improved in the time interval between lactate measurement and eligibility assessment. Lactate measurements more than 4 hours prior to eligibility assessment should not normally be used.
* Hospital presentation within last 12 hours

Exclusion Criteria:

* >1500ml of intravenous fluid prior to screening
* Clinically judged to require immediate surgery (within one hour of eligibility assessment)
* Immediate (< 1 hour) requirement for central venous access
* Chronic renal replacement therapy
* Known allergy/adverse reaction to norepinephrine
* Palliation / end of life care (explicit decision by patient/family/carer in conjunction with clinical team that active treatment beyond symptomatic relief is not appropriate)
* Previous recruitment in the trial
* Patients with permanent incapacity
* Pregnancy. All women of childbearing potential (WoCBP) must have a negative urine or serum pregnancy test result completed as part of screening requirements.

WoCBP are defined as fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause.

* Other primary causes of shock (e.g. suspected cardiogenic shock, haemorrhagic shock, etc)
* History or evidence of any other medical, neurological or psychological condition that would expose the subject to an undue risk of a significant Adverse Effect as determined by the clinical judgement of the investigator
* Participation in other clinical trials of investigational medicinal products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1006 (Estimated)
Dates: Start 2022-10-11 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to determine whether early PVI (within 12 hours of admission) targeted to MAP of ≥65 mmHg improves clinical effectiveness in hospitalised adult patients with septic shock compared with usual care, in the first 48 hours. | 90 days post randomisation
  The primary objective is measured by the Primary outcome of 'Days Alive and Out of Hospital at 90 Days'.

SECONDARY OUTCOMES:
Accumulated Total Volume of IV fluid | 6,12, 24, 48 and 72 hours post randomisation
  Accumulated volume of IV fluid delivered in each arm - excluding fluid volumes less than 100ml
Lactate clearance from baseline | 6, 12, 24, 48 & 72 hours post randomisation
  Blood lactate value - arterial or venous
Total Dose of Norepinephrine | 6, 12, 24, 48 and 72 hours post randomisation
  Total dose of norepinephrine delivered by any route (peripheral or central) at each timepoint
Proportion of patients who receive vasopressors | 6, 12, 24 and 48 hours after recruitment to the control arm
  Proportion of patients recruited to control arm who receive any vasopressor (norepinephrine, vasopressin, metarminol, epinephrine) at each time point
Proportion of patients who require central venous access | 24 and 48 hours post randomisation
  Decision to treat based on treating clinician judgement
Proportion of patients developing acute kidney injury | During the first 72 hours post randomisation
  Acute kidney injury in line with the (p) RIFLE (paediatric Risk, Injury, Failure, Loss, End stage renal disease, AKIN (Acute kidney injury network) or KDIGO (Kidney Disease: Improving Global Outcomes) definitions by using any of the following criteria
  * a rise in serum creatinine of 26 micromol/litre or greater within 48 hours
  * a 50% or greater rise in serum creatinine known or presumed to have occurred within the past 7 days
  * a fall in urine output to less than 0.5 ml/kg/hour for more than 6 hours in adults
Proportion of patients receiving parenteral corticosteroid | 24, 48 & 72 hours post randomisation
  defined as new prescription of parenteral corticosteroid
Length of hospital stay for index admission | up to hospital discharge
  index hospital admission ends when the patient is discharged from the facility providing definitive treatment for the episode of sepsis leading to inclusion in the study
Proportion of participants needing renal replacement therapy during index hospital admission | index admission
  decision to treat based on treating clinician judgement; participants who receive new renal replacement therapy; participants with chronic renal replacement initiated prior to the index admission will not be eligible to meet this endpoint
Proportion of participants needing non-invasive ventilation during index hospital admission | index admission
  decision to treat based on treating clinician judgement; defined as admissions receiving mask/hood CPAP or mask/hood BiPAP or non-invasive ventilation; admissions receiving CPAP via a tracheostomy
Proportion of participants needing advanced respiratory support (ICNARC definition) | index admission
  decision to treat based on treating clinician judgement; Patients who receive one or more of the following: A. Patients who receive invasive mechanical ventilation via endotracheal or tracheostomy tube, except those intubated solely for a procedure and extubated within 24 hours B. BiPAP (bilevel positive airway pressure) applied via a trans-laryngeal tracheal tube or applied via a tracheostomy C. CPAP (continuous positive airway pressure) via a translaryngeal tune of applied via a tracheostomy D. extracorporeal respiratory support
Total dose of other vasopressor | 6, 12, 24, 48, 72 hours post randomisation
  Total dose of other vasopressors delivered by any route (peripheral or central) at each timepoint
All-cause mortality during index hospital admission and at 30 and 90 days | index admission and at 30 & 90 days post randomisation
  All-cause mortality during index hospital admission and at 30 & 90 days post randomisation
Readmission, post initial hospital discharge, in first 30 days and 90 days post randomisation | 30 & 90 days post randomisation
  Re-admission to an acute healthcare facility in the first 30 & 90 days post randomisation, following a discharge from the index hospital admission to the participants care setting in the community. This includes planned and unplanned admissions. For both readmission outcomes, an acute care facility is any acute care hospital, emergency department admission >24 hours, critical care area or short stay admission or observation area.
Proportion of participants admitted to and length of stay in critical care (level 2 or 3) during index hospital admission | During Index Hospital Admission
  Proportion of participants admitted to and length of stay in critical care (level 2 or 3) during index hospital admission
Discharge Diagnosis | At initial Index Hospital Discharge & at any subsequent hospital discharges following any re-admissions (post Initial Index Hospital Discharge) 90 days post randomisation.
  Main diagnosis for index hospital admission, and all subsequent re-admissions
HRQoL | Baseline, 30 & 90 Days Post randomisation
  Derived from EQ-5D-5L index values

OTHER OUTCOMES:
Patient Centred Outcome | 30 days post randomisation
  organ support free days at 30 days
Protocol Adherence | 48 hours post randomisation
  Proportion of patients who have PVI discontinued for non-clinical reasons after recruitment to intervention arm
Protocol Adherence | 48 hours post randomisation
  Proportion of patients in control arm who receive PVI
Organ Dysfunction Score | Baseline Only (0 hours)
  Organ dysfunction score (SOFA) calculated at Baseline
Proportion of patients developing vasopressor extravasation | 72 hours post randomisation
  Proportion of patients developing vasopressor extravasation during first 72 hours
Proportion of patients developing pulmonary oedema | index admission
  Proportion of patients developing pulmonary oedema during index hospital admission

CONTACTS AND LOCATIONS:
Locations (25):
- United Kingdom (25):
  - Aintree University Hospital, Aintree
  - Royal Blackburn Hospital, Blackburn
  - Fairfield General Hospital, Bury
  - Addenbrookes Hospital, Cambridge, Cambridge
  - Royal Derby Hospital, Derby
  - Royal Infirmary of Edinburgh, Edinburgh
  - Victoria Hospital, Fife Keith
  - Glasgow Royal Infirmary, Glasgow
  - Queen Elizabeth University Hospital, Glasgow
  - Hull Royal Infirmary, Hull
  - Kettering General, Kettering
  - University Hospital Crosshouse, Kilmarnock
  - University Hospital Monklands, Lanark
  - Leicester Royal Infirmary, Leicester
  - Royal Liverpool University Hospital, Liverpool
  - Newham University Hospital, London
  - Royal London Hospital, London
  - St George's, London
  - University Hospital Lewisham, London
  - John Radcliffe Hospital, Oxford
  - Royal Alexandra Hospital, Paisley
  - Peterborough City Hospital, Peterborough
  - Royal Berkshire Hospital, Reading
  - Queens Hospital Barking, Romford
  - Salford Royal, Salford

IPD SHARING:
Plan to Share IPD: No
to be confirmed